CLINICAL TRIAL: NCT01521221
Title: Assessment of Hand-grip in the Prevention of Postural Orthostatic Hypotension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-08-AM-462-CTIL
Record Dates: First submitted 2011-08-15; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Experimental): Patients with autonomic failure.
  Interventions: Other: Hand grip maneuver
- Healthy subjects (Experimental): Control group
  Interventions: Other: Hand grip maneuver

INTERVENTIONS:
Other: Hand grip maneuver — Hand grip on blood pressue cuff slightly inflated at 50-70% of maximal force for 1 minute

SUMMARY:
The study is aimed to assess the efficacy of hand-grip in preventing orthostatic hypotension in 20 patients diagnosed with autonomic failure. Five healthy subjects will be studied for comparison. The investigators will evaluate the subjects while on tilt table for 10 minutes and than while mounted from lying down to 70 degrees for additional 10 minutes. Blood pressure, heart rate and symptoms will be continuously measured. First study will evaluate the blood pressure changes. Second measure will include hand-grip maneuver 1 minute before the erect positon. Trans cranial Doppler will assess the intracranial blood flow during the position changes.

DETAILED DESCRIPTION:
Study 1:

10 minutes lying on the tilt table. Performing TCD study at 10 minutes. Raising the tilt table to 70 degrees. Performing TCD study 5 minutes after tilting. Measuring blood pressure and symptoms for 10 minutes. Returning the tilt bed to supine position.

Study 2. in continue with study 1:

10 minutes lying on the tilt table. Performing TCD study at 10 minutes. Performing hand-grip at 50-70% grip force for 1 minute Raising the tilt table to 70 degrees. Performing TCD study 5 minutes after tilting. Measuring blood pressure and symptoms for 10 minutes. Returning the tilt bed to supine position.

ELIGIBILITY:
Inclusion Criteria:

* Man or women
* 18 years of age or older
* Diagnosed with orthostatic hypotension due to Parkinson's disease, multiple system atrophy or pure autonomic failure
* Orthostatic hypotension is not due to drugs, any heart disorder, anemia or dehydration

Exclusion Criteria:

* Pregnant or breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in orthostatic blood fall after tilting with and without hand grip. | 10 minutes after tilting the subjects.
  Patients will be tilted to 70 degrees twice. Hand grip maneuver will be performed 1 minute before the second tilt study and the differences in blood pressure changes [baseline-end tilt (mmHg)] will be compared between the two studies and to those obtained from a healthy control group.

SECONDARY OUTCOMES:
Change in the intracranial blood flow after tilting with and without hand grip. | 10 minutes after tilting.
  Intracranial blood flow will be evaluated by transcranial doppler at baseline and after tilting. Differences will be compared [peak systolic flow (PSW) cm/sec], after tilting with and without prior hand grip and in comparison to tilting a control group.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Mosek, MD, Principal Investigator — Deputy Chief, the Department of Neurology, Sourasky Medical Center
Locations (1):
- Movement disorders unit, the Department of Neurology, Sourasky Medical Center, Tel Aviv, Israel